CLINICAL TRIAL: NCT02602145
Title: Optimal Stent Selection for the Femoropopliteal Artery
Acronym: SFA
Status: Terminated | Type: Observational
Why Stopped: Study team did not maintain IRB approval
Sponsor: University of Nebraska (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0386-14-FB; 5R01HL125736-05 (NIH)
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Femoropopliteal Stenting
Keywords: femoral; popliteal; stent; modeling; flexion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peripheral artery disease patients: Patients with peripheral artery disease who were treated with a stent as part of their standard of care. Patients who meet the inclusion criteria (i.e. already have a stent in their femoropopliteal artery) will be consented after their endovascular repair, and those who choose to participate in the study will be followed for 6-12 months. During the follow-up, a post-operative contrast-enhanced CTA of the lower extremities will be obtained to assess for restenosis.
  Interventions: Other: follow-up CTA

INTERVENTIONS:
Other: follow-up CTA — All patients will receive PAD stents as their normal standard of care determined by their treating physician. If the patient would decide to enroll in the study, we will perform a post-operative contrast-enhanced CTA of the lower extremities at 6-12 months after stenting.

SUMMARY:
Angioplasty and stenting for atherosclerotic occlusive disease in the arteries supplying the legs (Peripheral Arterial Disease, PAD) is the most common endovascular procedure outside of the heart, but carries the highest rate of reconstruction failure. The underlying reasons for these poor results are not completely clear, but the main arterial segment within the leg, the femoropopliteal artery, appears to be significantly different from other peripheral arteries because the Superficial Femoral Artery (SFA) and Popliteal Artery (PA) that comprise the femoropopliteal artery (FPA) segment, undergo large deformations during flexion of the limb. We propose to build mathematical models of human FPAs repaired with several frequently used PAD stents. These mathematical models would be able to assess the mechanical stress in the stented SFA and PA associated with limb flexion and predict disease recurrence for arteries with different patient and lesion characteristics. Results of model predictions will be validated in patients with PAD stents who have received these stents as part of their standard of care.

DETAILED DESCRIPTION:
This is an observational study of PAD patients that have already received SFA and PA stents as part of their standard of care.

The purpose of this study is to determine the effects of Peripheral Artery Disease (PAD) stenting on the femoropopliteal artery. This will be achieved through the following Specific Aims:

Aim 1. Evaluate pre-operative lower extremity CTAs of patients with PAD and determine the baseline arterial geometry and lesion characteristics.

Aim 2. Evaluate the results of intraoperative angiography and blood pressure measurements proximal and distal to the stent.

Aim 3. After stenting perform post-operative lower extremity CTA and assess the amount of in-stent restenosis and changes to the arterial geometry.

We propose to build mathematical models of human femoropopliteal arteries repaired with several of the most commonly used PAD stents and assess the mechanical stress associated with limb flexion. These models will aim at predicting disease recurrence for arteries with different patient and lesion characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for participating in this study are patients with severe PAD who have:

  1. endovascular repair of their femoropopliteal artery
  2. standard pre-operative contrast-enhanced thin-section CTA of the lower extremities
  3. intraoperative angiograms and blood pressure measurements proximal and distal to the stent during the endovascular repair
  4. no aneurysmal disease of the target femoropopliteal artery
  5. no prior open or endovascular repair of the target femoropopliteal artery (patients with re-interventions are not eligible)
  6. at least 2 out of 3 patent crural outflow vessels
  7. life expectancy >6 months
  8. no iodinated contrast allergy
  9. creatinine less than 1.6 g/dL (unless on chronic dialysis, dialysis patients are eligible)
  10. no orthopedic prostheses in the region of interest
  11. ability to comply with 6-12-month follow-up contrast enhanced thin-section CTA

Exclusion Criteria:

1. no endovascular repair of the femoropopliteal artery
2. endovascular or open re-intervention in the target limb
3. no pre-operative thin-section contrast-enhanced CTA of the target limb
4. no intraoperative angiogram or blood pressure measurements proximal and distal to the stent
5. aneurysmal disease of the target femoropopliteal artery
6. less than 2 patent crural outflow vessels
7. life expectancy ≤ 6 months
8. iodinated contrast allergy
9. orthopedic prosthesis in the region of interest
10. creatinine greater than 1.6 g/dL (unless dialysis patient, chronic dialysis patients are eligible)
11. inability to comply with 6-12-month contrast-enhanced CTA follow-up requirement
12. patient belongs to vulnerable population, i.e. pregnant women, prisoners, institutionalized individuals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe peripheral artery disease already treated with a stent.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Radius of the femoropopliteal artery lumen | 6-12 months
  Radius of the femoropopliteal artery lumen will be measured using follow-up CTA to assess narrowing of the artery after stent implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Jason MacTaggart, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States